CLINICAL TRIAL: NCT05748990
Title: Does Abnormal Insulin Action in the Brain Underlie Cognitive and Metabolic Dysfunction in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 154-2020
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Healthy
Keywords: schizophrenia; insulin; glucose; brain; PET; FDG; antipsychotic-naive; 18-fluorodeoxyglucose; intranasal insulin
MeSH Terms: conditions — Schizophrenia; Insulin Resistance | interventions — Insulin Lispro; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: In a single-blind crossover design, participants will undergo an [18F]-FDG PET scan on 2 separate occasions separated by 4-7 days. One of the PET scans will be following intranasal placebo (saline) and the other will follow an intranasal insulin challenge (160 IU). The scans will be conducted in a randomized counterbalanced order across participants to account for exposure to antipsychotics between the two scans.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schizophrenia Group (Experimental): Insulin (160IU) or placebo is administered intranasally 15 minutes prior to the PET scan.
  Interventions: Drug: Intranasal insulin; Drug: Placebo
- Healthy Control Group (Experimental): Insulin (160 IU) or placebo is administered intranasally 15 minutes prior to the PET scan.
  Interventions: Drug: Intranasal insulin; Drug: Placebo

INTERVENTIONS:
Drug: Intranasal insulin — 160 IU insulin (Humalog) is administered intranasally using a metered spray bottle 15 minutes prior to the PET scan.
  Other Names: Humalog
Drug: Placebo — 0.9% saline is administered intranasally using a metered spray bottle 15 minutes prior to the PET scan.
  Other Names: saline

SUMMARY:
Cognitive impairment (such as challenges in thinking and memory) is a core aspect of schizophrenia (SCZ), contributing to disability and poor functional outcomes. Additionally, almost half of the patients with SCZ are obese, the prevalence of type 2 diabetes is 3-6 times higher, and life expectancy is lower by 15-20 years compared to the general population. This is relevant as metabolic syndrome and diabetes are both associated with worse cognition among SCZ patients. Recent work studying the relationships between metabolic health and cognition has encouraged a new way of thinking about SCZ as both a metabolic and cognitive disorder. Brain insulin is involved in several processes relevant to SCZ, and abnormal brain insulin action may help explain both cognitive and metabolic abnormalities in patients with SCZ, but this has not been examined previously. Glucose uptake in several brain regions relevant to SCZ has been shown to be partially dependent on insulin. Therefore, in this study, the researchers will measure glucose uptake in the brain using an 18F-fluorodeoxyglucose ([18F]-FDG) positron emission tomography (PET) scan after an intranasal insulin stimulus, and will compare this measure between patients with SCZ and healthy controls.

DETAILED DESCRIPTION:
i) Schizophrenia and cognition: Cognitive impairment is a core aspect of schizophrenia (SCZ), contributing to disability and poor functional outcomes. Antipsychotics reduce positive symptoms but there are no currently approved treatments for cognitive impairment, creating a large unmet need.

ii) Schizophrenia and metabolic dysfunction: Patients with SCZ also have exceedingly high rates of metabolic comorbidity. Almost half of patients are obese and the prevalence of type 2 diabetes is 3-9 fold higher than the general population. Patients with SCZ die on average 15-20 years earlier than the general population from cardiovascular disease. Thus, metabolic health represents another large unmet need.

iii) Association between cognitive and metabolic dysfunction: These two domains of dysfunction interact in an additive manner to worsen outcomes. Metabolic syndrome and diabetes are both associated with worse cognition among SCZ patients. Recent knowledge elucidating the interactions between metabolic health, cognition, and functioning have encouraged a reconceptualization of SCZ as both a metabolic and cognitive disorder, prompting search for treatment strategies that address abnormalities in both these aspects.

iv) Brain insulin as a unifying link: There has been recent recognition that insulin plays an important role in the brain. Brain insulin is implicated in several processes relevant to SCZ. Abnormal brain insulin action may help explain both cognitive and metabolic aberrations in patients with SCZ. Moreover, it is now clear that glucose uptake in the brain is partially dependent on insulin in brain regions relevant to SCZ, such as the hippocampus, hypothalamus, and striatum.

v) Evidence and promise in SCZ: There is preliminary evidence to suggest that brain insulin resistance is associated with worse cognition. A magnetic resonance spectroscopy (1H-MRS) study found higher brain glucose and lower glucose utilization in SCZ patients, suggesting brain insulin resistance, that were associated with memory impairment. Initial intervention studies using intranasal insulin have not been successful, likely because resistance to insulin in the brain prevents any benefits of intranasal insulin from accruing. However, this has not been conclusively demonstrated. This study seeks to answer this question directly.

vi) Role of 18-fluorodeoxyglucose ([18F]-FDG)-positron emission tomography (PET): 1H-MRS is an indirect and imprecise measure of glucose in the brain (it combines intra- and extracellular glucose). This is also true for other MRI based measures, which have recently been employed to indirectly study insulin action in the brain. Currently, there are no PET ligands able to reliably quantify insulin or its receptors in the brain. However, using [18F]-FDG PET, it is possible to measure differences in glucose uptake, with and without an insulin challenge, into insulin sensitive regions of the brain (e.g. hippocampus and striatum). This can serve as a surrogate marker of brain insulin action. This principle has already been used successfully in rodents and healthy humans, and offers a more direct method of quantifying brain insulin action.

In this study, [18F]-FDG PET will be employed to examine whether abnormal brain insulin action is a feature of SCZ. The study examines young SCZ patients. Insulin (160 IU; shown to be safe and effective previously) will be delivered intranasally as it has been shown to be reliable method of delivering insulin to the brain.

Primary hypothesis: SCZ patients will have reduced [18F]-FDG uptake, in response to an intranasal insulin challenge, compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

i) Experimental group (participants with a diagnosis of schizophrenia spectrum disorder):

1. 17-45 years
2. both sexes;
3. Patients with first-episode schizophrenia spectrum illness: Primary DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, brief psychotic disorder, psychotic disorder NOS, major depressive disorder with psychotic symptoms, bipolar I disorder, and bipolar II disorder, OR substance-induced psychosis, and antipsychotic treatment for schizophrenia, schizoaffective disorder, or other specified schizophrenia spectrum, other psychotic disorder, major depressive disorder with psychotic symptoms, bipolar I disorder, and bipolar II. (Diagnosis willbe confirmed via CAMH chart review).
4. BMI under or equal to 27

ii) Control group (healthy controls):

1. 17-45 years of age
2. sex-,
3. hand dominance -and
4. body mass index (BMI)-matched
5. Absence of DSM-5 diagnosis other than a specific phobia according to MINI

Exclusion Criteria:

1. moderate or severe substance use according to MINI (per PI discretion in the case of moderate alcohol or cannabis use)
2. prediabetes, diabetes, or evidence of impaired glucose tolerance on screening OGTT
3. acute suicidal risk
4. use of weight, lipid, antidiabetic or blood pressure reducing agents
5. liver or kidney disease
6. pregnancy
7. nursing
8. pacemakers
9. metallic cardiac valves
10. magnetic material such as surgical clips, implanted electronic infusion pumps or any other conditions that would preclude the MRI scan
11. clinically significant claustrophobia (determined from MRI screening form; significance evaluated as per QI's discretion).
12. history of head trauma resulting in loss of consciousness > 30 minutes that required medical attention;
13. size of head, neck, precluding to fit in the MRI or PET scanners
14. weight over 350lbs (limit for MRI scanner bed)
15. unstable physical illness
16. significant neurological disorder including a seizure disorder;
17. Received maximum allowed radiation in the past 12 months (20 mSv)
18. Completed more than 6 PET scans/ lifetime, that, together with the PET scanning procedures under this protocol will bring the total number of PET scans to more than the allowed/lifetime (8 PET scans per lifetime). These limits are set by the Centre for Addiction and Mental Health Brain Health Imaging Centre Guideline.
19. clinically relevant abnormality observed in medical history,
20. current intake of any medication that may interfere with participation in the study or may confound the results of PET imaging (e.g. anti-diabetic medication).
21. Disorders of coagulation, blood or ongoing use of anticoagulant medication

Control group: Exclusionary criteria are as listed above for participants, in addition to:

1) First degree family member with primary psychotic disorder.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
[18F]-FDG brain uptake | Scan duration is ~90 minutes
  Change in [18F]-FDG uptake in striatum and hippocampus is measured in response to intranasal insulin challenge or placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No